CLINICAL TRIAL: NCT07152535
Title: Multi-omics Monitoring of Dynamic Evolution in Esophageal Squamous Cell Carcinoma: PKU-ESCC-Monitor
Acronym: PKU-ESCC
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PKU-ESCC-0604; LGH2025236 (Other: Peking University Cancer Hospital)
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC)
Keywords: ESCC; Multi-omics; ctDNA; Immunotherapy; Neoadjuvant Therapy; Prospective Cohort; Biomarkers
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Tumor biopsy before neoadjuvant/first-line therapy; surgical specimens and adjacent tissue from transthoracic esophagectomy; archived FFPE slides (3-5 μm, 5-8 slides when fresh tissue is unavailable); serial blood for ctDNA and cytokines (e.g., IL-6/IL-8). All specimens are obtained from routine clinical care with consent and retained for DNA analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Peri-operative ESCC Cohort: Patients with histologically confirmed ESCC who complete standard neoadjuvant therapy and undergo transthoracic esophagectomy. Study assigns no treatment; care is per treating physicians. Study procedures include collection of tumor tissue/surgical specimens or archived FFPE slides and serial blood for ctDNA/cytokines, plus prospective follow-up of clinical outcomes.
- Advanced ESCC First-line Immunotherapy Cohort: Patients with unresectable/advanced ESCC receiving standard-of-care first-line immunotherapy at participating centers. No assigned intervention by the study; all treatments are per routine practice. Study procedures include tumor biopsy or archived FFPE slides and serial blood for ctDNA/cytokines, with prospective follow-up for responses and survival.

SUMMARY:
This prospective observational study (PKU-ESCC-Monitor) aims to characterize the dynamic evolution of esophageal squamous cell carcinoma (ESCC) using integrated multi-omics, including tissue genomics, ctDNA, imaging features, immune profiling and microbiome. Two cohorts will be followed: a peri-operative cohort after standard neoadjuvant therapy and surgery, and an advanced cohort receiving first-line immunotherapy. Clinical outcomes (DFS/PFS/OS) and biomarker dynamics will be analyzed to improve risk stratification and response prediction.

DETAILED DESCRIPTION:
The study integrates clinical data with multi-omics (tumor tissue, surgical specimens, archived FFPE slides where applicable, serial blood for ctDNA and cytokines such as IL-6/IL-8, and exploratory immune/microbiome assessments). Patients are followed monthly or per routine visits up to 36-60 months. Analyses include RECIST 1.1-based responses (ORR, DCR, TTR, DOR), survival endpoints, and biomarker-clinical modeling to delineate ESCC evolutionary patterns and treatment response.

ELIGIBILITY:
Inclusion Criteria:

Peri-operative cohort:

1. Age ≥18 and <80 years; ECOG 0-1.
2. Histologically confirmed ESCC.
3. Completed standard neoadjuvant therapy and planned/underwent 4.transthoracic esophagectomy with routine surgical specimens available.

5.Able to provide clinical course/outcomes and comply with follow-up at participating sites.

Advanced first-line immunotherapy cohort:

1. Age ≥18 and <80 years; ECOG 0-1.
2. Histologically confirmed ESCC, or highly suspected by endoscopy/imaging when surgery is not feasible.
3. No prior systemic anti-cancer therapy for advanced disease; archived FFPE slides (3-5 µm, 5-8 slides) acceptable if fresh tissue unavailable.
4. Able to provide clinical information and comply with follow-up.

Exclusion Criteria:

1. Prior anti-cancer therapy (except standard neoadjuvant therapy in the peri-operative cohort).
2. Other malignancy within 5 years (exceptions: non-melanoma skin cancer, in-situ melanoma, in-situ cervical cancer).
3. Inadequate clinical information.
4. Known infection with HIV, HBV, HCV, or syphilis.
5. Pre-operative imaging indicates insufficient tumor tissue (no visible target region) for study procedures.
6. Any condition deemed by investigators to make the patient unsuitable.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (18-79 years) with histologically confirmed esophageal squamous cell carcinoma (ESCC) treated at Peking University Cancer Hospital and participating centers in China. Two prospective cohorts: (1) peri-operative patients who complete standard neoadjuvant therapy and undergo transthoracic esophagectomy; (2) unresectable/advanced ESCC receiving standard-of-care first-line immunotherapy. ECOG 0-1. Tumor tissue (biopsy or surgical; archived FFPE slides acceptable if fresh tissue is unavailable) and serial blood are collected for multi-omics analyses. Key exclusions include prior systemic therapy for advanced disease (except neoadjuvant in the peri-operative cohort), other active malignancies within 5 years (allowing non-melanoma skin and in-situ cervical cancer), inadequate clinical information, or investigator-assessed unsuitability.
Sampling Method: Non-Probability Sample
Enrollment: 255 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) | up to 60 months
  peri-operative cohort; time from study registration to first ESCC recurrence or death from any cause; patients alive without recurrence are censored at last contact.
Progression-Free Survival (PFS) | up to 36 months
  advanced cohort;time from start of first-line therapy to first documented disease progression per RECIST 1.1 or death.
Overall Survival (OS) | up to 60 months
  time from study registration to death from any cause.

SECONDARY OUTCOMES:
Time to Response (TTR) | up to 60 months
  time from study registration to first ESCC recurrence or death from any cause; patients alive without recurrence are censored at last contact.
Objective Response Rate (ORR) | best overall response up to 24 months; proportion with CR/PR by RECIST 1.1.
  up to 24 months
Disease Control Rate (DCR) | up to 24 months; proportion with CR/PR/SD by RECIST 1.1.
  up to 24 months
Biomarker Analyses | baseline to 36-60 months
  exploratory associations for PD-L1, HER2, EGFR, ctDNA dynamics, IL-6/IL-8 and other immune/microbiome markers with outcomes.

IPD SHARING:
Plan to Share IPD: Undecided